CLINICAL TRIAL: NCT05666167
Title: Expanding Exercise Programming for Veterans Through Telehealth (CDA 22-066)
Brief Title: Expanding Exercise Programming for Veterans Through Telehealth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CDX 22-008
Record Dates: First submitted 2022-11-17; First posted 2022-12-27 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Arthritis
Keywords: osteoarthritis; exercise maintenance; telehealth; group exercise; text messaging
MeSH Terms: conditions — Arthritis; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Initiation and Maintenance with Text Messaging and Booster Sessions (Experimental): Participants receive 3 months of group telehealth exercise initiation plus text messaging followed by 6 months of text messaging plus monthly group telehealth exercise booster sessions.
  Interventions: Behavioral: Group Telehealth Exercise Sessions with text messaging plus booster sessions
- Exercise Initiation and Maintenance with Text Messaging alone (Active Comparator): Participants receive 3 months of group telehealth exercise initiation plus text messaging followed by 6 months of text messaging alone.
  Interventions: Behavioral: Group Telehealth Exercise Sessions with text messaging plus booster sessions

INTERVENTIONS:
Behavioral: Group Telehealth Exercise Sessions with text messaging plus booster sessions — Participants receive 3 months of group telehealth exercise initiation plus text messaging followed by 6 months of text messaging plus monthly group telehealth exercise booster sessions.

SUMMARY:
The goal of this study is to evaluate the acceptability and feasibility of a group telehealth exercise program for Veterans with lower extremity osteoarthritis (OA). Methods: This is a randomized pilot trial where Veterans (n=50) receive a group telehealth exercise program (3 months), followed by an exercise maintenance phase (6 months) that includes either text messaging alone or text messaging plus group telehealth exercise booster sessions. The primary outcomes for this study are feasibility and acceptability of the intervention. Feasibility will be assessed through number and source of referrals, recruitment, and retention. Acceptability will be assessed through surveys and interviews for participants and providers addressing reasons for participation, satisfaction, perceived appropriateness, and overall experience containing Likert scales and both yes/no and open-ended questions. Exploratory outcomes, assessed at multiple time points during the course of the study, will measure changes in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and changes in performance measure and physical activity assessed remotely through individual telehealth sessions. Data will be collected at baseline, 3-, 6-, and 9-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of symptomatic knee or hip OA
* Veterans at Eastern Colorado Healthcare System Primary Care Clinics with at least one VA visit within the past year
* physically inactive (add definition)

Exclusion Criteria:

* No telephone access
* hip or knee surgery or acute meniscus or anterior cruciate ligament tear in the past six months
* recent hospitalization for cardiovascular/cerebrovascular event
* serious mental health condition or behavioral issues precluding participating in group exercise
* terminal illness
* motor neuron diseases
* severely impaired hearing, vision, or speech
* non-English speaking
* current participation in another OA or exercise intervention or lifestyle change study
* other self-reported or study team/primary care physician deemed health condition that would prohibit participation in the study
* no primary care physician visit in past 12 months
* pregnant women
* insufficient internet connectivity to participate in group telehealth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Referrals | 3 months
  The number of referrals made by providers, through chart review, and the number of self-referrals by Veterans will be collected as a measure of feasibility.
Number of sessions attended | 3 months
  The number of sessions attended as a percentage of the number offered will be gathered as a measure of feasibility and acceptability.
Recruitment | 3 months
  The goal is that 50% of eligible provider and self-referrals and 25% of chart review referrals will participate in the program as a measure of success.

SECONDARY OUTCOMES:
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Scores | Baseline, 3 months, 6 months, and 9 months.
  Changes in lower extremity pain (5 items), stiffness (2 items), and function (17 items) assessed using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scale scores. Each item is scored on a Likert scale ranging from 0 to 4 (none, mild, moderate, severe, and extreme). Scores range from 0-96 and higher scores are generally associated with worse outcomes.

OTHER OUTCOMES:
Change in 30-second chair stand test | Baseline, 3 months, 9 months
  Number of times participant can rise from sitting in a chair in 30 seconds. Higher scores indicate higher function.
Change in 2-minute Step Test | baseline, 3 months, 9 months
  The number of steps in place (right knee to midpoint of upper leg = 1 step) in 2 minutes. Higher scores indicate higher function.
Change in Arm Curls | Baseline, 3 months, 9 months
  The number of curls performed in 30 seconds. Higher scores indicate higher function.
Change in Accelerometry Data | Baseline, 3 months, 6 months, 9 months
  Gathered using an ActiGraph worn on wrist for 7 consecutive days. Specifically step changes in step counts. Larger increases indicate increased physical activity.
Change in Number of Steps assessed by Pedometer | Baseline, 3 months, 6 months, 9 months
  Daily steps recorded by Veteran in AnnieApp text message reply and in daily exercise logs. Larger increases indicate increased physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Abbate, MD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No